CLINICAL TRIAL: NCT05974293
Title: A Phase IIb Study of the Safety and Efficacy of Nabiximols in Subjects With Spasticity Due to Neuromyelitis Optica Spectrum Disorders: A Double-blind, Randomized, Placebo-Controlled, Crossover Study
Brief Title: A Phase IIb Study of Nabiximols for Spasticity Due to Neuromyelitis Optica Spectrum Disorders
Acronym: SENS-NMO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was withdrawn.
Sponsor: Michael, Levy M.D.,Ph.D. (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Michael, Levy M.D.,Ph.D., Associate Professor of Neurology at Massachusetts General Hospital, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023P002959
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: NMO Spectrum Disorder; Spasticity, Muscle
Keywords: Neuromyelitis Optica Spectrum Disorders; Nabiximols; Cannabinoid; Sativex
MeSH Terms: conditions — Neuromyelitis Optica; Muscle Spasticity; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: This is a phase II, single-site, double-blind, randomized, placebo-controlled 2 by 2 crossover clinical trial designed to evaluate the efficacy of nabiximols compared to placebo for the treatment of NMOSD-related spasticity.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nabiximols, then Placebo (Experimental): During Period 1, participants receive daily nabiximols spray, delivered by a pump action oromucosal spray. The first 2 weeks of Period 1 are the titration period with participants following pre-specified uptitration schedule, until they reach their individualized optimum daily dosage, with a maximum of 12 daily sprays. Following these 2 weeks, they continue the optimum dose for 4 weeks. Then, they undergo a 2-week washout period, and then, enter Period 2 where they receive the matched placebo spray and again undergo a 2-week titration period, and a 4-week consistent daily dosage period.
  Interventions: Drug: Nabiximols; Drug: Placebo
- Placebo, then Nabiximols (Experimental): During Period 1, participants receive daily matched placebo spray, delivered by a pump action oromucosal spray. The first 2 weeks of Period 1 are the titration period with participants following pre-specified uptitration schedule, until they reach their individualized optimum daily dosage, with a maximum of 12 daily sprays. Following these 2 weeks, they continue the optimum dose for 4 weeks. Then, they undergo a 2-week washout period, and then, enter Period 2 where they receive the active nabiximols spray and again undergo a 2-week titration period, and a 4-week consistent daily dosage period.
  Interventions: Drug: Nabiximols; Drug: Placebo

INTERVENTIONS:
Drug: Nabiximols — Nabiximols is is a yellow-brown oromucosal spray solution containing 27 mg/mL of THC and 25 mg/mL of CBD.
  Other Names: Sativex
Drug: Placebo — The placebo is a matching oromucosal spray that is identical to the investigational study product in terms of packaging, labelling, schedule of administration, dosing instructions, and appearance.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of nabiximols, a cannabinoid spray, for the treatment of moderate to severe spasticity in adult patients with AQP4-IgG positive and antibody-negative NMOSD. The main question it aims to answer is whether treatment with nabiximols improves patient-reported spasticity ratings compared to treatment with a placebo. This trial will also answer whether nabiximols impact pain, spasm frequency, mood, walking ability, and sleep. Participants will be mailed the treatments and placebo treatments, and will be asked to complete study visits and questionnaires remotely. There is also an optional sub-study that involves in-person visits with ultrasound imaging and in-person neurologic exams.

DETAILED DESCRIPTION:
Patients with NMOSD often have medication-resistant and severe spasticity due to longitudinally extensive spinal cord lesions. Existing treatments are limited by their efficacy and tolerability. Cannabinoids have been shown to quantitatively improve spasticity in mouse models of neuroinflammation, and nabiximols, a cannabinoid-based oromucosal spray, have demonstrated efficacy for medication-resistant spasticity in multiple sclerosis. However, no studies have as yet explored the use of nabiximols specifically in NMOSD, and there is a significant unmet need for new symptomatic treatments in this patient population. The goal of this study is to evaluate the safety and efficacy of nabiximols spray, for the treatment of moderate to severe spasticity in adult patients with AQP4-IgG positive and seronegative NMOSD. This study is designed as a phase IIb, single-site, double-blind, randomized, placebo-controlled 2x2 crossover clinical trial, with a 2-week washout period between treatment periods. After randomization, each participant enters into Period 1, which begins with a 2-week dose escalation period with a pre-defined dose escalation scheme, followed by a 4-week stable treatment period. After completion of Period 1, all participants have a 2-week washout period and then enter Period 2, where they again complete a 2-week dose escalation period and 4-week constant treatment period. The patient-reported 0-10 numeric rating scale for spasticity (NRS-S) is the primary outcome measure. All key study procedures are performed virtually, including a weekly electronic study diary, additional weekly surveys, and 8 virtual video-based study visits including a screening visit and safety follow up visit. Additional optional in-person assessments of spasticity (neurologic exam, modified Ashworth Scale and muscle ultrasound elastography) will be performed for a selection of local participants. In total, the study has a 20-week duration per participant, from the screening visit to the final study completion for safety follow-up visit, including 12 weeks of on-treatment time.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of NMOSD, meeting the International Panel for NMO Diagnosis (IPND) NMOSD criteria (Appendix 1), including NMOSD with AQP4-IgG, and NMOSD without AQP4-IgG
* Aged between 18 years or older, at the time of signing the informed consent
* Willing and able to give informed consent and to participate in all study procedures
* Moderate to severe spasticity, as defined by a score of > 3 on the 0-10 numerical rating scale for spasticity (NRS-S) at the time of screening
* Reports NMOSD-related spasticity symptoms ongoing for at least 6 months
* Spasticity is determined to be causally related to an NMOSD attack in the opinion of the investigator
* No relapses, and otherwise stable disease (i.e. no significant recovery from relapse or other change in disability) for at least 6 months, in the opinion of the investigator
* Anti-spasticity regimen, if on medications, maintained at a stable dose for the 30 days prior to enrollment without adequate relief of spasticity symptoms.
* Willing to maintain a stable dose of non-study-related anti-spasticity medication for the duration of the study, barring significant changes to their medical condition.
* Willing to allow his or her primary care doctor and primary neurologist, if appropriate, to be notified of participation in the study.
* Documentation of negative MOG-IgG, if diagnosis is NMOSD without AQP4-IgG positive status. Participant with presumptive diagnosis of NMOSD without AQP4-IgG and no prior MOG IgG testing can have MOG testing sent, and be eligible for participation if this is negative.
* For women of childbearing potential: participants who are not lactating, not pregnant, and not planning to become pregnant in the next 8 months and who agree to remain abstinent (refrain from heterosexual intercourse) or use adequate contraception during the treatment period and for at least 3 months after the final dose of nabiximols.
* For males with partners who are females of childbearing potential: participants who agree to remain abstinent (refrain from heterosexual intercourse) or use adequate contraception during the treatment period and for at least 3 months after the final dose of nabiximols.
* Able to use the necessary electronic applications (either via smartphone, tablet, or desktop) and has an email address.

Exclusion Criteria:

* Consumption of cannabis herb or other cannabinoid-based drugs within 30 days prior to study entry.
* Unwillingness to abstain from consumption of cannabis herb or other cannabinoid-based drugs for the duration of the study.
* Known or suspected hypersensitivity or adverse reaction (including psychiatric adverse reactions) to cannabinoids or cannabinoid products, ethanol, peppermint oil or propylene glycol.
* Currently receiving a prohibited medication and unwilling or unable to stop for the duration of the study. Prohibited medications include: CYP3A4 inhibitors: clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, verapamil, etc.; CYP3A4 inducers: rifampicin, phenobarbital, phenytoin, St. John's Wort. Of note, the CYP3A4 inducer carbamazepine is permitted, but a stable dosage must be maintained throughout the study (no as needed dosing permitted). Other prohibited medications: regular levodopa (Sinemet, Sinemet Plus, Levodopa, L-dopa, Madopar, Benserazide), sildenafil (Viagra), fentanyl, or antiarrhythmic medications.
* Receipt of an investigational medicinal product or participation in a therapeutic clinical trial within 30 days prior to the initial visit
* Received a Botulinum Toxin injection within four months prior to the screening visit or unwillingness to stop receiving Botulinum Toxin injections for the relief of spasticity for the duration of the study.
* Personal medical history of schizophrenia, severe personality disorders, other major psychotic disorders, or other major psychiatric disorders other than depression and anxiety.
* Family history in 1st degree relatives of schizophrenia or other psychotic disorders.
* Hospitalization for depression or anxiety within the 2 years prior to the screening visit.
* A documented history of attempted suicide or suicidal ideation of category 4 or 5 according to the Columbia Suicide Severity Rating Scale (C-SSRS) screening, OR if in the Investigator's judgment, the participant is at risk for a suicide attempt.
* Known or suspected history of a substance use disorder or heavy alcohol consumption excluding tobacco use disorder or cannabis use not meeting criteria for cannabis use disorder.
* History of myocardial infarction or clinically significant ischemic heart disease, arrhythmias (other than well controlled atrial fibrillation), poorly controlled hypertension or severe heart failure. .
* Significant renal or hepatic impairment, either in the opinion of the investigator, or by the following laboratory screening values: AST or ALT > 2 × upper limit of normal (ULN); Total bilirubin > 2 × ULN (unless due to Gilbert's syndrome); BUN > 2 × upper limit of normal (ULN)
* History of epilepsy or recurrent seizures.
* Concomitant disease or disorder that has symptoms of spasticity, and that in the opinion of the Investigator may influence the study outcome and endpoint assessment.
* Any other significant medical or psychiatric condition which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study or the participant's ability to participate in the study.
* Scheduled elective surgery or other procedures which require general anesthesia during the study period.
* Intention to donate blood during the study.
* Intention to travel internationally during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-12-31 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean Numeric Rating Scale - Spasticity (NRS-S) scores from pre-treatment to post-treatment | Baseline; Up to week 18
  Numeric Rating Scale - Spasticity (NRS-S) score is a 0-10 point, patient-reported scale indicating spasticity severity.

SECONDARY OUTCOMES:
Proportion of participants with NRS-S response corresponding to a minimal clinically important difference (MCID) (>18% difference) from pre-treatment to post-treatment | Baseline; Up to week 18
  Numeric Rating Scale - Spasticity (NRS-S) score is a 0-10 point, patient-reported, single item scale indicating spasticity severity.
Proportion of participants with NRS-S response corresponding to a clinically important difference (CID) (>30% difference) from pre-treatment to post-treatment | Baseline; Up to week 18
  Numeric Rating Scale - Spasticity (NRS-S) score is a 0-10 point, patient-reported scale indicating spasticity severity.
Change in Penn Spasm Frequency Scale (PSFS) score from pre-treatment to post-treatment | Baseline; Up to week 18
  The Penn Spasm Frequency Scale (PSFS) is a 2-item patient-reported scale indicating spasm frequency and severity
Change in mean PROMIS NRS v1.0 - Pain Intensity 3a scores from pre-treatment to post-treatment | Baseline; Up to week 18
  The PROMIS NRS v1.0 - Pain Intensity 3a form is a 3-item patient-reported scale indicating worst pain, average pain, and current pain in the prior week
Change in mean PROMIS SF v1.1 - Pain Interference 8a scores from pre-treatment to post-treatment | Baseline; Up to week 18
  The PROMIS SF v1.1-Pain Interference 8a form is an 8-item scale indicating the degree to which pain interferes with functioning
Change in mean Multiple Sclerosis Spasticity Scale - 88 (MSSS-88) sub-scale 2 (pain and discomfort) scores from pre-treatment to post-treatment | Baseline; Up to week 18
  The Multiple Sclerosis Spasticity Scale - 88 (MSSS-88) form sub-scale 2 (pain and discomfort) is a 9-item patient-reported scale indicating the impact of spasticity on pain and discomfort
Change in Floodlight-5 U-Turn Test (5-UTT) from pre-treatment to post-treatment | Baseline; Up to week 18
  The Floodlight-5 U-Turn Test (5-UTT) is a smartphone application-based test that evaluates ambulation, and specifically turn speed in seconds
Change in Floodlight-2 Minute Walk Test (2MWT) from pre-treatment to post-treatment | Baseline; Up to week 18
  The Floodlight-2 Minute Walk Test (2MWT) is is a smartphone application-based test that evaluates ambulation speed in seconds
Change in mean Multiple Sclerosis Spasticity Scale - 88 (MSSS-88) sub-scale 5 (walking) scores from pre-treatment to post-treatment | Baseline; Up to week 18
  The Multiple Sclerosis Spasticity Scale - 88 (MSSS-88) form sub-scale 2 (pain and discomfort) is a 10-item patient-reported scale indicating the impact of spasticity on walking
Change in PROMIS SF v1.0 - Sleep Disturbance 4A from pre-treatment to post-treatment | Baseline; Up to week 18
  The PROMIS SF v1.0 - Sleep Disruption 4A is a 4-item patient-reported scale indicating sleep quality
Change in Numeric Rating Scale-Sleep Disruption (NRS-SD) from pre-treatment to post-treatment | Baseline; Up to week 18
  The Numeric Rating Scale-Sleep Disruption (NRS-SD) is a single-item 0-10 scale where participants can indicate the degree to which spasticity impacts sleep
Proportion of participants reporting 'very much improved,' 'much improved,' and 'slightly improved' symptoms in the Global Impression of Change (GIC) by subject (SGIC) scores from pre-treatment to post-treatment | Baseline; Up to week 18
  The Global Impression of Change (GIC) by subject (SGIC) is a 7-point, single-item scale indicating the direction and degree of change that participants experience
Change in Visual Analogue Scale - Quality of Life (VAS-QL) from pre-treatment to post-treatment | Baseline; Up to week 18
  The Visual Analogue Scale - Quality of Life (VAS-QL) is a 100mm visual analog scale ranging from 0 (very low) to 100 (very high) on which respondents record their perception of quality of life
Proportion of participants who are tolerant of treatment | Screening; Up to week 18
  Tolerance is defined as not discontinuing study drug and at least 50% compliance
Proportion of participants who are tolerant of treatment | Screening; Up to week 20
  Tolerance is defined as not discontinuing study drug and at least 50% compliance
Number of participants with treatment-emergent adverse events while on each treatment | Screening; Up to week 20
  Treatment-emergent adverse events will be tabulated for each arm during each study period and compared between treatment and placebo
Columbia-Suicide Severity Rating Scale (C-SSRS) Score at Screening and at each subsequent time-point with reference to the last assessment | Screening; Up to week 20
  The Columbia-Suicide Severity Rating Scale is assessment tool that evaluates suicidal ideation and behavior

OTHER OUTCOMES:
Change in mean Patient Health Questionnaire-8 (PHQ-8) scores from pre-treatment to post-treatment | Screening; Up to week 20
  The Patient Health Questionnaire-8 is an 8-item self-administered depression scale
Change in mean PROMIS SF v1.0 - Anxiety 4a scores from pre-treatment to post-treatment | Screening; Up to week 20
  The PROMIS SF v1.0 - Anxiety 4a scale is a 4-item self-administered anxiety questionnaire
Change in mean Floodlight-Pinching Test (PT) scores from pre-treatment to post-treatment | Screening; Up to week 18
  The Floodlight-Pinching Test (PT) is a smartphone application-based test assessing hand and arm function
Change in mean Floodlight-Draw a Shape Test (DaS) scores from pre-treatment to post-treatment | Screening; Up to week 18
  The Floodlight-Draw a Shape Test (DaS) is a smartphone application-based test assessing hand and arm function
Change in mean Floodlight-e-Symbol Digit Modalities Test (eSDMT) scores from pre-treatment to post-treatment | Screening; Up to week 18
  The Floodlight-Draw a Shape Test (DaS) is a smartphone application-based test assessing cognition
Change in Lower Limb Muscle Tone-6 (LLMT-6) scores as measured by the modified Ashworth Scale scores from pre-treatment to post-treatment | Screening; Up to week 18
  LLMT-6 is defined as the average of the 6 individual Modified Ashworth Scale (MAS) transformed scores of knee flexors, knee extensors, and plantar flexors on both sides of the body
Change in muscle shear wave speed from pre-treatment to post-treatment | Screening; Up to week 18
  Muscle shear wave speed is measured using shear wave elastography, an ultrasound-based technique to assess muscle stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Massachusetts General Hospital; Anastasia Vishnevetsky, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No specific plan to share individual participant data with other researchers.